CLINICAL TRIAL: NCT00757510
Title: Congenital Heart Disease Research Registry
Acronym: CHDRR
Status: Terminated | Type: Observational
Why Stopped: Insufficient funding
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Associate Professor, Emory University
Other Study IDs: IRB00006304
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and serum collected from Registry subjects will be cryopreserved for potential future genetic and/or protein-based studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Congenital heart disease: All subjects will have known or suspected congenital heart disease

SUMMARY:
The Congenital Heart Disease Research Registry (CHDRR) is a program dedicated to understanding the etiology and improving the treatment of Congenital Heart Disease (CHD). This Registry will act as a central coordinating center for recruiting subjects with CHD and will provide infrastructure and guidelines for researchers studying the causes and treatment of CHD. Investigators working directly with the Registry will have access to biological, demographic and phenotype data from a significant pool of participants with CHD.

DETAILED DESCRIPTION:
The Registry will recruit participants from either new referrals for evaluation of potential CHD or from patients who are being followed within the Children's Healthcare of Atlanta Sibley Heart Center or Emory University Adult Congenital Heart Clinic with specific diagnoses and therapy. Participants will provide a biological sample (blood), demographic data, medical records and phenotypic data, and assessment data. These data will be stored in a secure database accessible only to investigators with research projects that have been approved by the IRB and by the executive committee of the CHDRR. The executive committee of the CHDRR will contain at least one member from each of the following: Sibley Heart Center, Emory Pediatric Cardiac Surgery Division, and Emory-Egleston Children's Research Center. This committee will meet quarterly to discuss patient enrollment, patient safety issues, and data integrity. They will also meet as needed to discuss any applications for sample utilization and study publications.

Blood and serum collected from Registry members will be cryopreserved for potential future genetic and/or protein-based studies. Note that no genotyping or analysis will be done by the Registry. The data collected is meant to give future researchers a base of information to establish eligibility for their specific studies. It is the goal of the Registry to work with researchers to gain IRB approval either to access scrubbed data or to contact Registry members for potential enrollment in any IRB-approved studies that would require access to private healthcare information (PHI).

Approved investigators can use the Registry database in two ways: 1) to query and extract data that have been scrubbed of identifiers, utilizing bar-code linked, de-identified blood or serum; and 2) to identify Registry members who are eligible for specific research projects requiring further patient contact. In the latter application, the investigators will identify potential participants via the scrubbed data, but will not have access to personal information during the initial identification process. The Registry research coordinator will then contact the identified Registry members, explain the study, and request consent to give their contact information to the investigator. The investigator will then contact consenting, eligible members using their IRB approved, project-specific protocol. In both applications, IRB approval will be required before the Registry database will be accessed or samples released for study. Further, investigators will be required to report participation outcomes of eligible Registry members to the Registry research coordinator. The Registry research coordinator will track participation/refusal/non-participation of each Registry member who is identified and contacted for additional research projects.

ELIGIBILITY:
Inclusion Criteria:

* All patients suspected or diagnosed with congenital heart disease receiving care at Children's Healthcare of Atlanta or Emory University Adult Congenital Heart Clinic and willing to sign informed consent.

Exclusion Criteria:

* Not referred or diagnosed with CHD
* No informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suspected or diagnosed with congenital heart disease receiving care at Children's Healthcare of Atlanta or Emory University Adult Congenital Heart Clinic
Sampling Method: Non-Probability Sample
Enrollment: 861 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
There is no outcome measure. This is a data, blood and serum collection only to provide a base for future studies | We will be collecting samples for a minimum of 40 years.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Kirshbom, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] McElhinney DB, Geiger E, Blinder J, Benson DW, Goldmuntz E. NKX2.5 mutations in patients with congenital heart disease. J Am Coll Cardiol. 2003 Nov 5;42(9):1650-5. doi: 10.1016/j.jacc.2003.05.004. PMID 14607454
- [Background] Lambrechts D, Devriendt K, Driscoll DA, Goldmuntz E, Gewillig M, Vlietinck R, Collen D, Carmeliet P. Low expression VEGF haplotype increases the risk for tetralogy of Fallot: a family based association study. J Med Genet. 2005 Jun;42(6):519-22. doi: 10.1136/jmg.2004.026443. No abstract available. PMID 15937089
- [Background] Goldmuntz E. The genetic contribution to congenital heart disease. Pediatr Clin North Am. 2004 Dec;51(6):1721-37, x. doi: 10.1016/j.pcl.2004.08.006. PMID 15561182
- [Background] Walther T, Schubert A, Falk V, Binner C, Walther C, Doll N, Fabricius A, Dhein S, Gummert J, Mohr FW. Left ventricular reverse remodeling after surgical therapy for aortic stenosis: correlation to Renin-Angiotensin system gene expression. Circulation. 2002 Sep 24;106(12 Suppl 1):I23-6. PMID 12354704
- [Background] Kerstann KF, Feingold E, Freeman SB, Bean LJ, Pyatt R, Tinker S, Jewel AH, Capone G, Sherman SL. Linkage disequilibrium mapping in trisomic populations: analytical approaches and an application to congenital heart defects in Down syndrome. Genet Epidemiol. 2004 Nov;27(3):240-51. doi: 10.1002/gepi.20019. PMID 15389927